CLINICAL TRIAL: NCT00328081
Title: State of Obesity Care in Canada Evaluation Registry An Observational Study of Clinical Care of Patients With Obesity
Brief Title: State of Obesity Care in Canada Evaluation Registry
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left the institution
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Abbott (Industry)
Organization: McMaster University (Other)
Other Study IDs: SOCCER
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Obesity; Morbid Obesity
Keywords: Obesity; Weight gain; Anti-obesity medication; Anti-obesity management strategies; Body Weight
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Gain; Body Weight

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to see whether care gap(s) exist in the management of obesity and its related conditions in obese patients seen by primary care physicians and specialists. The study will also look at whether there is a compliance and adherence gap that exists in patients prescribed medication for obesity management.

DETAILED DESCRIPTION:
Obesity currently affects over 15% of the adult population in Canada. The economic burden associated with obesity is estimated at $4.3 billion or 2.2% of the total health care costs in Canada. Despite increasing recognition as a public health problem, clinical management of obese patients in Canada has received little attention. This study will collect information on the current status, characteristics and management of subjects with obesity. The design of the study will mirror real-life management of these subjects.There are three goals in this study: the primary goal is to document appropriate obesity management strategies aimed at reducing and maintaining a healthy body weight by participating primary care physicians and specialists. The second goal is to explore factors that determine patients compliance and adherence to anti-obesity medication when prescribed. Obesity management is currently not a priority in tertiary care centres in Canada. An exception being the Bariatric Clinic located at McMaster University, which is one of the few academic centers dedicated to obesity management in Canada. The primary goal of the Bariatric Clinic Substudy is to evaluate the management, compliance and adherence of patients seen at a tertiary care obesity clinic compared to those of primary care physicians and specialists.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and is able to provide informed consent
* Has not been enrolled in this study at an earlier office visit; and
* Provides signed informed consent
* BMI > = 27 kg/m

Exclusion Criteria:

* Participation in a clinical trial
* Hospitalized patient
* Subject expected to have difficulties to come back at follow-up visits
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1906 (Actual)
Dates: Start 2006-05; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arya M Sharma, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - Cardiovascular Obesity Research and Management, Hamilton, Ontario, Canada